CLINICAL TRIAL: NCT00961779
Title: A Phase I, Double-Blind, Randomized, Dose Escalation Study to Assess the Safety, Tolerability and PK of NNZ-2566 in Healthy Females, When Administered as a Loading Dose (10-Min), and as a Loading Dose Followed by a Maintenance Dose (72-Hr).
Brief Title: Safety Study of NNZ-2566 in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neu-2566-HV-004
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — trofinetide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Normal saline infusion) (Placebo Comparator)
  Interventions: Drug: Placebo
- NNZ-2566 (Experimental): NNZ-2566 reconstituted in bicarbonate buffer and normal saline. 6/8 subjects in each cohort (5 cohort in total) to receive NNZ-2566 experimental treatment.
  Interventions: Drug: NNZ-2566

INTERVENTIONS:
Drug: NNZ-2566 — Glycyl-L-2-Methylprolyl-L-Glutamic Acid (NNZ-2566) supplied as a lyophilized powder (2g in 50mL vials) for reconstitution with bicarbonate buffer and normal saline.
  Other Names: Experimental name: NNZ-2566
  Arms: NNZ-2566
Drug: Placebo — Normal saline infusion
  Other Names: Sodium Chloride 0.9% Injection
  Arms: Placebo (Normal saline infusion)

SUMMARY:
The purpose of this study is to obtain evidence of the safety of NNZ-2566 in healthy female volunteers and to determine the pharmacokinetics (PK) of NNZ-2566 in healthy female volunteers.

DETAILED DESCRIPTION:
To obtain evidence of the safety of NNZ-2566 in healthy female volunteers, compared to placebo when administered as a 10 minute intravenous (i.v.) bolus infusion, and when administered as a 10-minute bolus infusion immediately followed by a continuous 72-hour maintenance infusion.

To determine the blood pharmacokinetics (PK) of an intravenous dose of NNZ-2566 in healthy female volunteers when administered as a 10-minute bolus infusion, and when administered as a 10-minute bolus followed by a continuous 72-hour maintenance infusion.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 years and 50 years (inclusive).
* Females only.
* Weight 50 to 105 kg
* BMI of 18 to 30 kg/m2.
* General Health: Healthy, determined by a medical history with particular attention to:

  * a drug history identifying any known drug allergies and the presence of drug abuse;
  * any chronic use of medication; and
  * a thorough review of body systems. This will also be determined by having no clinically significant abnormal findings on physical examination, which includes an electrocardiogram (ECG), which in the opinion of the Investigator would jeopardize the safety of the subject or impact on the validity of the study results.
* Venous Access: Volunteers with adequate venous access in their left and right arm to allow collection of blood samples and drug administration.
* Language: Fluent in the English language.
* Informed Consent: Have voluntarily given written informed consent to participate in this study.

Exclusion Criteria:

* Pregnant and lactating females are excluded from participating in the study.
* History of allergy and/or hypersensitivity to any of the stated ingredients of the formulations.
* History of clinically significant gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease or hematological disorders.
* Any history of asthma during the last 10 years.
* A creatinine clearance of less than 75 mL/min.
* Any predisposing condition that might interfere with the absorption, distribution, metabolism, and/or excretion of the investigational product.
* History of abnormal bleeding tendencies or thrombophlebitis unrelated to venepuncture or intravenous cannulation.
* History of Hepatitis B, a positive test for Hepatitis B surface antigen, a history of Hepatitis C, a positive test for Hepatitis C antibody, a history of HIV infection or demonstration of HIV antibodies.
* Pregnancy.
* Any evidence of organ dysfunction, or any clinically significant clinical laboratory value, including a liver function test (LFT) > 1.5 x upper limit of normal (ULN).
* Difficulty abstaining from alcohol during the 48 hours prior to dose administration and until completion of blood sampling at exit assessment.
* History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit, or positive urine drug screen for drugs of abuse.
* Difficulty in abstaining from any prescription medications for 14 days prior to dose administration and for the duration of the study.
* Difficulty in abstaining from over-the-counter (OTC) medications or herbal supplements for 14 days prior to dose administration and for the duration of the study, (with the exception of occasional analgesia, vitamin and other nutrient supplement use, at the discretion of the Investigator).
* Difficulty in abstaining from food and/or beverages that contain caffeine or other xanthines, (e.g., coffee, tea, cola and chocolate) during the 24 hours prior to dose administration and whilst confined at the clinical study facility.
* History of any psychiatric illness which may impair the ability to provide written informed consent.
* Poor protocol compliers or those unlikely to attend.
* Receipt of any drug as part of a research study within 30 days of initial dose administration in this study.
* Standard blood donation (usually 550 mL) within the 12-week period before dose administration.
* Unusual dietary habits and excessive or unusual vitamin intakes.
* Vaccination or immunizations within 30 days of initial dose administration.
* QT/QTc Exclusions i.e., a marked baseline prolongation of corrected QT interval > 450 ms in two ECGs, or a history of risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | Through to Day 7 post end of study drug infusion or until resolved

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Wilson, MB ChB, PhD, Study Director — Neuren Pharmaceuticals Ltd
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia